CLINICAL TRIAL: NCT05418179
Title: Effect of Probiotic Supplementation on Fecal Microbiota, Nutritional Status, Metabolic and Inflammatory Parameters in Patients With Type 2 Diabetes Mellitus: Study Protocol for a Triple-blind Controlled Randomized Clinical Trial
Brief Title: Effect of Probiotic Supplementation on Fecal Microbiota, Nutritional Status, Metabolic and Inflammatory Parameters in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Santa Catarina (Other)
Responsible Party: Principal Investigator, Erasmo Benicio Santos de Moraes Trindade, Professor, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UFSC_2021
Record Dates: First submitted 2022-06-05; First posted 2022-06-14 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study participants and researchers were masked over consumption and distribution of supplementation, respectively.
  Laboratory technicians who performed the blood collection were also masked as to the distribution of supplementation.
  Supplements and placebo were pre-packaged by the supplier in opaque and closed sachets with randomization codes, being identical in physical appearance, taste and color. Supplement identification codes were only disclosed by the supplier after statistical analysis of study data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Maltodextrin (1 capsule/day)
  Interventions: Dietary Supplement: Placebo
- Probiotic (Active Comparator): Probiotic (Bifidobacterium animalis subsp. Lactis, Bifidobacterium breve, Bifidobacterium longum, Lactobacillus gasseri, Lactobacillus casei, Lactobacillus rhamnosus) - 1 capsule/day
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic (Bifidobacterium animalis subsp. Lactis, Bifidobacterium breve, Bifidobacterium longum, Lactobacillus gasseri, Lactobacillus casei, Lactobacillus rhamnosus) - 1 capsule/day
  Arms: Probiotic
Dietary Supplement: Placebo — Maltodextrin (1 capsule/day)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of probiotic supplementation on fecal microbiota, nutritional status, metabolic and inflammatory parameters in patients with type 2 diabetes mellitus.

Study hypothesis: Supplementation of multispecies probiotic (Bifidobacterium Lactis, B. brebe, B. longum, Lactobacillus gasseri, L. casei, L. rhamnosus) during 12 weeks improves the the fecal microbiota composition and promotes reduction of plasma/serum levels of acute phase proteins, cytokines, metabolic and anthropometric parameters in individuals with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of multispecies probiotic supplementation (specifically designed for the present study) on fecal microbiota, nutritional status, metabolic and inflammatory parameters in patients with type 2 diabetes mellitus (T2DM).

Adult individuals (35 to 75 years old) of both sexes with T2DM (diagnosed at least 1 year ago), body mass index from 25.00 kg/m² to 39.99 kg/m², glycated hemoglobin ≤ 9.0% and using metformin will be invited to participate in this randomized, placebo-controlled, triple-blind study.

The participants will be randomized into two groups: G1 - probiotic group and G2 - control group (placebo).

The study will consist of two experimental time points: M0 - baseline and start of supplementation; M1 - after 12 weeks of the first outpatient visit and start of supplementation.

In the two experimental moments, individual fecal samples will be obtained for analysis of the fecal microbiota; The metabolic parameters will be assessed by determination of circulating levels of SCFA, FFA, insulin, fasting glucose and glycated hemoglobin, HOMA-IR; Total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides; the inflammatory response will be assessed by determination of plasma indicadors (LPS, Adiponectina, IL-10, IL-1, IL-6, TNF- α, Leptina, Resistina) ; besides the evaluation of indicators of nutritional status (bone densitometry with body composition and anthropometric measurements).

The primary endpoint will be the fecal microbiota composition, SCFA concentrations and the inflammatory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age from 35 to 75 years old;
* Individuals diagnosed with type 2 diabetes mellitus (at least 1 year ago);
* Body mass index from 25.00 kg/m² to 39.99 kg/m²;
* Glycated hemoglobin ≤ 9.0% ;
* Using metformin, combined or not with other antidiabetic drugs

Exclusion Criteria:

* Previous bowel diseases (inflammatory bowel disease and irritable bowel syndrome); or previous gastrointestinal surgery (eg, colectomy, gastrectomy)
* Intolerances and ∕ or food allergies with a previous medical diagnosis (eg lactose intolerance or celiac disease);
* Glomerular filtration rate <30 ml/min/1.73m²; inflammatory diseases and immunodeficiencies;
* Diagnosis of autonomic neuropathy with gastrointestinal involvement such as: diabetic gastroparesis, diabetic enteropathy (diarrhea) or colonic hypomotility (constipation);
* Hospital admission and/or use of anti-inflammatory drugs (non-hormonal and corticosteroids) up to 1 month before the study; and ∕or use of antibiotics up to 3 months before the study;
* Regular use of laxatives, opioid narcotic analgesics or appetite suppressants;
* Current or previous use (up to 1 month) of prebiotics, probiotics, symbiotics or products enriched with these food supplements;
* Intolerance to prebiotics, probiotics or symbiotics;
* Pregnant or breastfeeding;
* Follow-up of a diet, guided by a nutritionist, for weight loss or gain up to 1 month before the study or current follow-up of unusual diets (eg vegetarian, macrobiotic, paleolithic);
* Alcohol consumption (> 1 drink/day or 14g of alcohol for women; >2 drinks/day or 28 grams of alcohol for men); use of illicit drugs and smokers;
* Change of lipid-lowering and/or antidiabetic drugs in the last 3 months

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-24 (Estimated)

PRIMARY OUTCOMES:
Fecal Microbiota | 12 weeks compared to baseline
  analysis method: 16s rRNA sequencing and bioinformatics analysis. Reported measure: taxonomic profiles of the microbial populations (operational taxonomic units / OTUs)
SCFA | 12 weeks compared to baseline
  Acetate, propionate, isobutyrate, butyrate and isovalerate (μmol/L)
Inflammatory parameters | 12 weeks compared to baseline
  Plasma LPS, adiponectin, leptin, resistin, IL-1, IL-6, IL-8, IL-10 and TNF-alpha concentrations (pg/mL)

SECONDARY OUTCOMES:
Fasting insulin | 12 weeks compared to baseline
  μUI/mL
fasting blood glucose | 12 weeks compared to baseline
  mg/dL
HOMA-IR | 12 weeks compared to baseline
  HOMA-IR = [fasting blood glucose (mmol) x fasting insulin (UI/ml)] ÷ 22,5
Glycated hemoglobin | 12 weeks compared to baseline
  percentage (%)
Free Fat Acids | 12 weeks compared to baseline
  µmol/L
Triglycerides | 12 weeks compared to baseline
  mg/dL.
Total cholesterol | 12 weeks compared to baseline
  mg/dL
LDL-c | 12 weeks compared to baseline
  (Friedewald equation) LDL-c = total colesterol - HDL-c - Triglicerídeos/5
  Reported measure: mg/dL
HDL-c | 12 weeks compared to baseline
  mg/dL
Bone densitometry | 12 weeks compared to baseline
  Dual X-ray Absorptiometry (DXA). Reported measure: T-score and Z-score
Body weight (kg) | 12 weeks compared to baseline
  kilograms
Waist circumference (cm) | 12 weeks compared to baseline
  centimeters (cm)
Body mass index (BMI) | 12 weeks compared to baseline
  In metric units: BMI (kg/m²) = weight (kg) ÷ height² (meters). Reported measure: kg/m².
Total Body Fat Percentage (%BF) | 12 weeks compared to baseline
  Dual X-ray Absorptiometry (DXA). Reported measure: Total Body Fat Percentage (%BF)
Fat Mass Index (FMI) | 12 weeks compared to baseline
  Dual X-ray Absorptiometry (DXA) - Fat Mass Index (FMI) - the total amount of fat (in kilograms) relative to the height (in meters²)
Total Body lean mass Percentage (%) | 12 weeks compared to baseline
  Dual X-ray Absorptiometry (DXA) - Total Body lean mass Percentage (%): The percent of the body that is not composed of fat.

CONTACTS AND LOCATIONS:
Locations (1):
- Polydoro Ernani de São Thiago University Hospital, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Undecided